CLINICAL TRIAL: NCT04549207
Title: A Randomised Trial Comparing Continuation or De-escalation of Bone Modifying Agents (BMA) in Patients Treated for Over 2 Years for Bone Metastases From Either Breast or Castration-resistant Prostate Cancer (REaCT-Hold BMA)
Brief Title: Comparing Continuation or De-escalation of Bone Modifying Agents (BMA) in Patients Treated for Over 2 Years for Bone Metastases From Either Breast or Castration-resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REaCT-Hold BMA
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Castration-resistant Prostate Cancer
Keywords: Bone modifying agents; BMA; Breast cancer; Castration-resistant prostate cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid; Denosumab; Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard BMA frequency (Active Comparator): Continue standard BMA frequency (every 4 or 12 weeks) as administered previously. If a change in BMA frequency (every 4 weeks to every 12 weeks OR every 12 weeks to every 4 weeks) was prescribed by the physician, this would still be considered on protocol treatment.
  Interventions: Drug: Bone modifying agent
- De-escalate BMA to once every 24 weeks (Active Comparator): Bone modifying agent once every 24 weeks.
  Interventions: Drug: Bone modifying agent

INTERVENTIONS:
Drug: Bone modifying agent — Use of bone modifying agent
  Other Names: Zoledronate; Denosumab; Pamidronate

SUMMARY:
The investigators propose to perform a pragmatic, multicenter, open-label, randomised clinical trial to demonstrate the efficacy and safety of either continuing or further de-escalating BMA after a minimum of two years of BMA treatment in patients with bone metastases from breast cancer and castration-resistant prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with either radiologically and/or histologically confirmed bone metastases from castrate resistant prostate cancer or breast cancer who are currently receiving BMA
* Patient has received BMA for 2 or more years counting from the first BMA dose for bone metastases
* Age 18 years or older
* Able to provide verbal consent

Exclusion Criteria:

* Definite contraindication for BMA
* History of, or current evidence of osteonecrosis of the jaw
* Radiotherapy or surgery to the bone planned within 4 weeks after randomization
* Current hypercalcemia defined as corrected serum calcium of > 3 mmol/L (from standard bloodwork completed within one month prior to treatment dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life scores | 48 weeks after randomization (one year of treatment)
  Health related quality of life (HR-QoL) scores measured by the European Organisation for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ)-C30 physical functioning subscale and the European Organisation for Research and Treatment of Cancer (EORTC)- Quality of Life Questionnaire (QLQ)- for patients with bone metastasis (BM)22 functional interference subscale. The EORTC-QLQ-C30 is an internationally accepted and validated tool in multiple large study cohorts capturing HR-QoL from a multi-dimensional and global perspective in oncology. EORTC-QLQ-BM22 has been validated for use specifically in bone metastases. They were developed in collaboration with patients, healthcare professionals and thorough review of the literature, and therefore important to all stakeholders; the scales are well-defined and easily measured, and HR-QoL is a relevant goal of care in the palliative care setting.

SECONDARY OUTCOMES:
Symptomatic Skeletal Event (SSE) | 2 years post-randomization
  Number of patients with one or more SSEs (defined as: use of radiotherapy to relieve skeletal symtoms, new symptomatic pathological bone fractures [vertebral or non-vertebral], spinal cord compression, tumour-related orthopedic surgical intervention, or hypercalcaemia] during trial period) up to 2 years post-randomization.
Time to development of Symptomatic Skeletal Event | 2 years post-randomization
  Defined from the date of randomization until the first date of patient experience an SSE. Any patient who does not experience an SSE will be censored on the last follow-up date and the patient can be confirmed as SSE-free (up to 2 years).
Symptomatic Skeletal Event-free survival | 2 years post-randomization
  SSE-free survival (composite of time to first SSE and time to death)
Skeletal morbidity | 2 years post-randomization
  Skeletal morbidity rate defined as ration of number of SSEs for each subject divided by the subject's time at risk in years.
Quality of life of cancer patients using the EORTC-QLQ-C30 | 48 weeks post-randomization
  Assess quality of life of cancer patients using the EORTC-QLQ-C30 (cancer patient specific questionnaire) at each time point, up to and including 48 weeks ("one year of treatment")
Quality of life of cancer patients using the EORTC-QLQ-BM22 | 48 weeks post-randomization
  Assess quality of life of cancer patients using the EORTC-QLQ-BM22 (patients with bone metastases specific questionnaire) at each time point, up to and including 48 weeks ("one year of treatment")
BMA-related toxicity rates | 2 years post-randomization
  BMA-related toxicity rates (up to 2 years) based on standard of care blood tests and clinical assessments
Incremental cost-effectiveness rations | 2 years post-randomization
  Defined as the difference in cost between two possible interventions, divided by the difference in their Quality Adjusted Life Year (QALY) gained.

OTHER OUTCOMES:
Frequency of subsequent de-escalation or discontinuation of BMAs | 2 years post-randomization
  In the continuation arm, frequency of subsequent de-escalation or discontinuation of BMAs
Frequency of restarting standard dosing BMA | 2 years post-randomization
  In the de-escalation arm, frequency of restarting standard dosing BMA (and the reasons for restarting)
Overall survival | 2 years post-randomization
  Overall survival during study duration

CONTACTS AND LOCATIONS:
Overall Officials: Terry Ng, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (5):
- Canada (5):
  - William Osler Health System, Brampton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario

REFERENCES:
- [Background] Ng TL, Tu MM, Ibrahim MFK, Basulaiman B, McGee SF, Srikanthan A, Fernandes R, Vandermeer L, Stober C, Sienkiewicz M, Jeong A, Saunders D, Awan AA, Hutton B, Clemons MJ. Long-term impact of bone-modifying agents for the treatment of bone metastases: a systematic review. Support Care Cancer. 2021 Feb;29(2):925-943. doi: 10.1007/s00520-020-05556-0. Epub 2020 Jun 13. PMID 32535678
- [Background] AlZahrani M, Clemons M, Vandermeer L, Sienkiewicz M, Awan AA, Hutton B, Pond GR, Ng TL. Real-world practice patterns and attitudes towards de-escalation of bone-modifying agents in patients with bone metastases from breast and prostate cancer: A physician survey. J Bone Oncol. 2020 Nov 10;26:100339. doi: 10.1016/j.jbo.2020.100339. eCollection 2021 Feb. PMID 33294318
- [Background] Alzahrani M, Clemons M, Sienkiewicz M, Shrem NS, McGee SF, Vandermeer L, Sehdev S, Savard MF, Awan A, Canil C, Hutton B, Pond G, Saunders D, Ng T. Perceptions around bone-modifying agent use in patients with bone metastases from breast and castration resistant prostate cancer: a patient survey. Support Care Cancer. 2021 Nov;29(11):6903-6912. doi: 10.1007/s00520-021-06238-1. Epub 2021 May 22. PMID 34023950
- See also: The Rethinking Clinical Trials (REaCT) website — https://react.ohri.ca/